CLINICAL TRIAL: NCT02950961
Title: Implementation of Tailored Collaborative Care For Women Veterans (CCWV) (QUE 15-272)
Brief Title: Collaborative Care for Women Veterans
Acronym: CCWV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-008
Record Dates: First submitted 2016-10-21; First posted 2016-11-01 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Depression; Stress Disorders, Post Traumatic
Keywords: Anxiety [F01.470.132]; Depression [F01.145.126.350]; Stress Disorders, Post-Traumatic [F03.950.750.500]; Primary Health Care [N04.590.233.727]; Mental Health [F02.418]; Patient Satisfaction [N05.300.150.600.630]; Patient Preference [N05.300.150.600.630.500]; Physicians, Primary Care [M01.526.485.810.800]; Physicians, Women [M01.526.485.810.820]; Health Behavior [F01.145.488]
MeSH Terms: conditions — Anxiety Disorders; Depression; Combat Disorders; Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Mixed Methods Implementation Evaluation (Other): The investigators used mixed methods to evaluate the implementation in two VA Women's Practice Based Research Network (PBRN) sites, describing services and patterns of care utilized by patients prior to seeing a care manager, and then 30, 60, 180, and 365 days post initiation of care with the care manager. Investigators also evaluated facilitators and barriers to implementation of this collaborative care model.
  Interventions: Behavioral: Collaborative Care for Women Veterans

INTERVENTIONS:
Behavioral: Collaborative Care for Women Veterans — This is a collaborative care model that focuses on identifying need for depression and/or anxiety care. Patients with possible anxiety and/or depression are referred to a care manager in primary care-mental health integration. The care manager then conducts a thorough assessment, offers the patient a variety of appropriate treatment options, and works with the patient to determine a care plan. One of the key options the investigators offered in this study is the Calm Tools for Living (CALM) intervention, which is focused on anxiety and which is rooted in patient preferences. Patients can choose web-based cognitive behavioral therapy (CBT) and/or pharmacologic treatment. In this study the investigators trained appropriate MH providers in CALM and studied the ways in which the intervention needs to be tailored to women Veterans.
  Other Names: Gender-Tailored Primary Care-Mental Health Integration

SUMMARY:
Implementation of Tailored Collaborative Care for Women Veterans (CCWV) was designed to enhance primary care-mental health integration for women Veterans by tailoring services to women Veterans' and providers' needs and providing an evidence-based intervention, Coordinated Anxiety Learning and Management, to address anxiety and depression in a patient-centered approach. CCWV was implemented in two of the Women's Health Practice-Based Research Network sites, with careful attention to local tailoring and adaptation to enhance the fit of the care model in varied local contexts.

DETAILED DESCRIPTION:
Background: Women Veterans are the fastest growing segment of Veterans Health Administration (VHA) users. This dramatic growth has created challenges for VHA. Gender disparities persist in cardiovascular (CV) and diabetes risk factor control, and rates of depression, anxiety, and mental health comorbidity are disproportionately high among women Veterans. Furthermore, a high rate of women Veterans' attrition from VA care, along with organizational barriers to care, substantiate that organizational changes are needed in order to engage and retain women Veteran VHA users in evidence-based, patient-centered care.

Objectives: The Enhancing Mental and Physical health of Women through Engagement and Retention (EMPOWER) QUERI addresses VHA Blueprint for Excellence Strategy 6, by advancing "personalized, proactive, patient-centered" care models, and Transformational Strategy 7.2.g by implementation of innovative care models in women Veterans' health care." The EMPOWER QUERI Program was designed to improve women Veterans' engagement and retention in evidence-based care for three high priority health conditions, i.e., prediabetes, cardiovascular, and mental health. To achieve this impact goal, the investigators proposed a cohesive portfolio of projects with the following aims: (1) To use an evidence-based implementation strategy that emphasizes local tailoring of care models, multilevel stakeholder engagement, and systematic evaluation of complex implementation processes in order to enrich organizational capacity for innovations in women Veterans' VHA health care; (2) To implement personalized, proactive, patient-centered innovations in VHA women's health that are acceptable, feasible, satisfactory, relevant, and effective for both providers and patients, thereby encouraging women Veterans' engagement and retention and sustainability of the innovations; and, (3) To generate implementation "playbooks" for the investigators' partners that are scalable and serve as guidance for future implementation of a broader array of evidence-based women's health programs and policy.

Methods: Three projects were conducted by an experienced multidisciplinary team. This trial pertains to "Implementation of Tailored Collaborative Care for Women Veterans," which evaluated implementation of an evidence-based collaborative care model tailored to enhance provider- and system-level capabilities to address women Veterans' anxiety and depression treatment needs, thereby improving organizational primary care-mental health integration (PC-MHI) effectiveness and women Veterans' engagement and retention in PC-MHI. This implementation research study used mixed methods implementation evaluation to investigate primary implementation outcomes of adoption, acceptability, feasibility, and reach. Multilevel stakeholder engagement was prioritized. Program-wide organizational-, provider-, and patient-level data was utilized to enhance synergy, productivity, and impact. Several implementation outcomes were assessed using qualitative methods and will be reported elsewhere (e.g. final report, manuscripts).These include Adoption of Care Model, Acceptability of Care Model, Feasibility of Care Model, and Satisfaction With Care Model.

As a coherent program of women's health implementation research and quality improvement, the EMPOWER QUERI constituted a major milestone in achieving Blueprint for Excellence (BPE) strategies and realizing women Veterans' engagement and, ultimately, empowerment in the VHA system.

ELIGIBILITY:
Inclusion Criteria

Patient Participants:

* Women VA patients with possible or confirmed anxiety and/or depression and/or PTSD

Provider Participants:

* VA staff in a primary care and/or mental health clinic

  * Note: gender based inclusion criteria did not apply to provider participants

Exclusion Criteria

Patient Participants:

* Male gender
* Cognitive impairment that would preclude completion of informed consent

Provider Participants:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women VA patients with possible or confirmed anxiety and/or depression and/or PTSD.
  Participant eligibility is based on self-representation of gender identity.
Enrollment: 153 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison B Hamilton, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Ariel J. Lang, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finley EP, Huynh AK, Farmer MM, Bean-Mayberry B, Moin T, Oishi SM, Moreau JL, Dyer KE, Lanham HJ, Leykum L, Hamilton AB. Periodic reflections: a method of guided discussions for documenting implementation phenomena. BMC Med Res Methodol. 2018 Nov 27;18(1):153. doi: 10.1186/s12874-018-0610-y. PMID 30482159
- [Derived] Hamilton AB, Farmer MM, Moin T, Finley EP, Lang AJ, Oishi SM, Huynh AK, Zuchowski J, Haskell SG, Bean-Mayberry B. Enhancing Mental and Physical Health of Women through Engagement and Retention (EMPOWER): a protocol for a program of research. Implement Sci. 2017 Nov 7;12(1):127. doi: 10.1186/s13012-017-0658-9. PMID 29116022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 patient participants; 30 provider participants
Period: Overall Study
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Started | 123
Completed | 116
Not Completed | 7
Not completed — Study had to stop due to COVID. | 7

BASELINE CHARACTERISTICS:
Population: 123 baseline patient participants
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (11.24695)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 30
  White | 62
  More than one race | 6
  Unknown or Not Reported | 11
number of mental health visits for the 30 days prior to care manager initiation [Count of Participants; unit: Participants] — Describing services and patterns of care utilized by patients for the 30 days prior to seeing a care manager.
  Participants
    1 visit | 48
    2 visits | 38
    3 visits | 18
    4 visits | 9
    5 visits | 4
    6 visits | 2
    0 visits | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Utilization of Services (30 Days)
Description: Change in utilization of services comparing utilization 30 days prior to 30 days post initiation of care with the care manager.
Time Frame: 30 days
Population: 7 participants are not included here due to COVID shut down.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 116
Participants
  utilization decreased | 53
  no change in utilization | 23
  utilization increased | 40

2. Primary Outcome: Change in Utilization of Services (60 Days)
Description: Change in utilization of services comparing utilization 60 days prior to 60 days post initiation of care with the care manager.
Time Frame: 60 days
Population: 7 participants are not included here due to COVID shut down.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 116
Participants
  utilization decreased | 40
  no change in utilization | 14
  utilization increased | 62

3. Primary Outcome: Change in Utilization of Services (180 Days)
Description: Change in utilization of services 180 days prior to 180 days post initiation of care with the care manager.
Time Frame: 180 days
Population: 7 participants are not included here due to COVID shut down.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 116
Participants
  utilization decreased | 29
  no change in utliization | 10
  utilization increased | 77

4. Primary Outcome: Change in Utilization of Services (365 Days)
Description: Change in utilization of services comparing utilization 365 days prior to 365 days post initiation of care with the care manager.
Time Frame: 365 days
Population: 7 participants are not included here due to COVID shut down.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 116
Participants
  utilization decreased | 28
  no change in utilization | 8
  utilization increased | 80

5. Primary Outcome: Change in Referrals
Description: Using the nonrandomized stepped wedge design, we will compare referrals to PC-MHI at baseline at each site, and compare to referrals throughout the 18-month implementation phase.
Time Frame: baseline, 18 months (implementation phase)
Population: It was pre-specified that a sample size of at least 260 patients at a minimum of 4 sites was required. With only 116 patients across 2 sites, the final numbers were not sufficient to fit the nonrandomized stepped wedge model. Therefore, data were not collected.
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

6. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: brief measure of global health: Patient-Reported Outcomes Measurement Information System (PROMIS)
Time Frame: 6 months
Population: The outcome measure was on a patient survey that had administration deferred due to IRB delays. This led to only 5 six-month follow up patient surveys completed at 1 site. The sample (N=5) is less than 5% of the overall study sample and not representative. Privacy issues due to the potentially identifiable nature of such a small sample restrict us from any reporting, as our sample does not meet the VA National Data Systems threshold for reporting aggregate data to protect confidentiality.
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

7. Primary Outcome: Overall Anxiety Severity and Impairment Scale (OASIS)
Description: brief measure of anxiety: Overall Anxiety Severity and Impairment Scale (OASIS)
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

8. Primary Outcome: Patient Health Questionnaire for Depression and Anxiety (PHQ-4)
Description: brief measure of depression: Patient Health Questionnaire for Depression and Anxiety (PHQ-4)
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

9. Primary Outcome: WHO Disability Assessment Schedule (WHODAS) Out Of Role Days Items
Description: brief measure of impact of disability on role functioning: WHO Disability Assessment Schedule (WHODAS) Out Of Role Days items
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

10. Primary Outcome: Global Rating of Satisfaction/Quality of Care
Description: brief measure of satisfaction and quality that we have used in several surveys of women Veteran VA patients
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

11. Primary Outcome: Altarum Consumer Engagement
Description: brief measure of patient engagement in care
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

12. Primary Outcome: Health Literacy (Chew et al. 2004)
Description: brief measure of health literacy: (Chew et al. 2004)
Time Frame: 6 months
Population: as for outcome 6
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: Adverse events were monitored only for patients who were enrolled in the survey and interview research components, but not for patients whose deidentified clinical data were used for this study.
Arm/Group | Arm 1: Mixed Methods Implementation Evaluation
All-Cause Mortality (participants affected / at risk) | 0/123
Serious Adverse Events (participants affected / at risk) | 0/123
Other Adverse Events (participants affected / at risk) | 0/123

LIMITATIONS AND CAVEATS:
Our implementation outcomes were assessed using qualitative methods

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02950961/Prot_SAP_000.pdf